CLINICAL TRIAL: NCT01534013
Title: Clinical Assessment of a Closed-loop Insulin Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13SM0363
Record Dates: First submitted 2012-01-30; First posted 2012-02-16 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Closed loop insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Closed-loop insulin delivery (Experimental): The closed loop device (bio-inspired artificial pancreas device, subcutaneous glucose monitor and insulin pump) will be applied to participants with type 1 diabetes
  Interventions: Device: The Imperial College Closed-Loop Insulin Delivery System
- Open-loop (Control visit) (Active Comparator): Subcutaneous glucose monitor and pump will be applied to participants with type 1 diabetes
  Interventions: Device: Open loop

INTERVENTIONS:
Device: The Imperial College Closed-Loop Insulin Delivery System — The Imperial College closed-loop insulin delivery system comprises 3 main components: the glucose sensor, the control algorithm and the insulin delivery system.
  Other Names: Closed-loop insulin delivery system; Artificial pancreas; Bio-inspired artificial pancreas
  Arms: Closed-loop insulin delivery
Device: Open loop — glucose sensor and pump
  Arms: Open-loop (Control visit)

SUMMARY:
The purpose of the study is to assess the safety and efficacy of the Imperial College closed loop insulin delivery system (artificial pancreas) in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
Background:

Type 1 diabetes is caused by antibodies attacking insulin-producing β-cells in the pancreas. Treatment is usually by regular insulin injections, informed by glucose measurements from fingerprick blood samples. However, injections do not mimic the normal behaviour of the β-cell and this leads to suboptimal blood glucose control and complications including kidney failure, blindness, nerve damage and heart disease. Aggressive treatment can help but may lead to potentially-dangerous low blood glucose levels (hypoglycaemia). Glucose control is measured by HbA1c (normal range 4 to 6%), a measure of the amount of haemoglobin exposed to glucose over a period of around 3 months.

Current regimens for treating Type 1 diabetes in clinical practice are mainly based on injections of subcutaneous insulin several times daily in dosages determined by intermittent blood glucose measurements. The DCCT (Diabetes Control and Complications Trial) demonstrated that intensive management using these principles reduced complications by 50-76%. This was at the expense of increased hypoglycaemia, especially at HbA1c levels <7.5%. In other studies, intensive management resulted in people spending 30% of the day with glucose values >10mM and >2 hours/day in hypoglycaemia, often at night.

A closed loop system provides the potential to improve HbA1c while avoiding hypoglycaemia. It requires continuous glucose measurement, a control device and a pump for insulin delivery. The subject has been extensively reviewed. Intelligent control devices have been developed by others, using the principles of feedback control or predictive modelling. These were initially cumbersome e.g. the 'biostator' but more recent systems have been miniaturised and are capable of achieving blood glucose control in the fasting state, when provided with an input of interstitial glucose levels. They have not yet proven robust, may be associated with hypoglycaemia and are not capable of achieving adequate post-prandial control nor of coping with intercurrent illness outside hospital environments.

This clinical trial protocol assesses the Imperial College closed loop insulin delivery system. The closed loop insulin delivery comprises 3 main components: the glucose sensor, the control algorithm and the insulin delivery system.

The glucose sensor that will be used throughout the clinical validation studies is a CE marked, MHRA approved device manufactured by Medtronic. It is a subcutaneous sensor which sits just under the skin and samples interstitial fluid using an enzyme electrode. A small voltage is applied across the sensor and a current is fed back to the sensor instrumentation. This current is proportional to the glucose concentration in interstitial fluid and is calibrated against blood glucose a minimum of 12 hourly.

The control algorithm is derived from physiological experiments carried out by other groups which have demonstrated how the beta cells in the pancreas produce insulin in people without diabetes. Utilising the data from these experiments it has been possible to implement the behaviour of the beta cell in software and we have used a simulator with 200 virtual patients to demonstrate the safety and efficacy of the software. The data from the simulator is attached to this application as an appendix. The simulator was developed from human data and takes into account sensor errors, sensor placement, route of insulin administration and meal-time glucose absorption. It has been approved by the FDA in the United States as a step in the pathway of developing an artificial pancreas and has been validated against human data. In the clinical validation device the control algorithm is implemented on a printed circuit board using a programmable micro-controller.

The insulin pump device used throughout the clinical validation is the Roche Accu-Check Combo Spirit. This is a CE marked MHRA approved device and will be supplied by Roche with capability for direct communication from the motor so that we can verify the pump is doing what the software commands and with a license to use the communications protocol for research purposes. This ensures safe communication between the control algorithm and the pump and provides a fail-safe to ensure that the pump motor is responding appropriately to the control algorithm.

Clinical validation of the closed loop insulin delivery device follows a path of incremental challenges to the algorithm and hardware, starting with a fasting basal study in advisory mode and progressing to ambulatory, meal studies in full closed loop.

The aim of this trial is to assess the safety and efficacy of the closed loop device by applying the technology to participants with type 1 diabetes in a variety of scenarios, starting with a fasting test and progressing to overnight control, mealtime control and, finally, an ambulatory test.

Brief outline of each of the 5 visits within the trial period:

* Visit 1: Screening including clinical examination, fasting blood tests, completion of diabetes quality of life questionnaire, continuous glucose monitor attached to subject
* Visit 2: Review of continuous glucose monitoring results after 5 days
* Visit 3: Short Duration Fasting Closed Loop (6 hours of closed-loop assessment)
* Visit 4: Long Duration/ Overnight Fasting Closed Loop and Standard Meal Challenge (13 hours of closed-loop assessment)
* Visit 5: 24 Hour Ambulatory Automatic Closed Loop

During visits 3-5 blood sampling for capillary glucose & ketones, venous glucose and insulin levels will take place every 15-30 minutes while the closed-loop insulin delivery system is running.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Type 1 diabetes confirmed on the basis of clinical features and a fasting c-peptide <200nmol/L
* Type 1 diabetes for greater than 1 year
* Continuous subcutaneous insulin infusion for greater than 6 months
* HbA1c < 8.5% (69mmol/mol)

Exclusion Criteria:

* Recurrent severe hypoglycaemia
* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials
* Have active malignancy or under investigation for malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Johnston, MBChB,PhD,FRCP, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, St Mary's Campus, London, United Kingdom

REFERENCES:
- [Background] Georgiou P, Toumazou C. A silicon pancreatic Beta cell for diabetes. IEEE Trans Biomed Circuits Syst. 2007 Mar;1(1):39-49. doi: 10.1109/TBCAS.2007.893178. PMID 23851519
- [Background] Georgiou P, Toumazou C. Towards an ultra low power chemically inspired electronic beta cell for diabetes. Circuits and Systems, 2006. ISCAS 2006. Proceedings. 2006 IEEE International Symposium on, p. 173, 2006.
- [Background] Ho M, Georgiou P, Singhal S, Oliver NS, Toumazou C. A bio-inspired closed loop insulin delivery based on the silicon pancreatic beta-cell. Circuits and Systems, 2008. ISCAS 2008. IEEE International Symposium on, pp. 1052-1055, 2008
- [Background] Oliver N, Georgiou P, Johnston D, Toumazou C. A benchtop closed-loop system controlled by a bio-inspired silicon implementation of the pancreatic beta cell. J Diabetes Sci Technol. 2009 Nov 1;3(6):1419-24. doi: 10.1177/193229680900300623. PMID 20144397
- [Background] Hovorka R. Continuous glucose monitoring and closed-loop systems. Diabet Med. 2006 Jan;23(1):1-12. doi: 10.1111/j.1464-5491.2005.01672.x. PMID 16409558
- [Background] Nathan D, Cleary P, Backlund J, Genuth S, Lachin J, Orchard T, Raskin R, Zinman B. Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes,
- [Background] Albisser AM, Leibel BS, Ewart TG, Davidovac Z, Botz CK, Zingg W. An artificial endocrine pancreas. Diabetes. 1974 May;23(5):389-96. doi: 10.2337/diab.23.5.389. No abstract available. PMID 4598089
- [Background] Schaller HC, Schaupp L, Bodenlenz M, Wilinska ME, Chassin LJ, Wach P, Vering T, Hovorka R, Pieber TR. On-line adaptive algorithm with glucose prediction capacity for subcutaneous closed loop control of glucose: evaluation under fasting conditions in patients with Type 1 diabetes. Diabet Med. 2006 Jan;23(1):90-3. doi: 10.1111/j.1464-5491.2006.01695.x. PMID 16409572
- [Background] Kovatchev BP, Breton M, Man CD, Cobelli C. In silico preclinical trials: a proof of concept in closed-loop control of type 1 diabetes. J Diabetes Sci Technol. 2009 Jan;3(1):44-55. doi: 10.1177/193229680900300106. PMID 19444330
- [Background] Thome-Duret V, Reach G, Gangnerau MN, Lemonnier F, Klein JC, Zhang Y, Hu Y, Wilson GS. Use of a subcutaneous glucose sensor to detect decreases in glucose concentration prior to observation in blood. Anal Chem. 1996 Nov 1;68(21):3822-6. doi: 10.1021/ac960069i. PMID 8914483
- [Derived] Reddy M, Herrero P, El Sharkawy M, Pesl P, Jugnee N, Thomson H, Pavitt D, Toumazou C, Johnston D, Georgiou P, Oliver N. Feasibility study of a bio-inspired artificial pancreas in adults with type 1 diabetes. Diabetes Technol Ther. 2014 Sep;16(9):550-7. doi: 10.1089/dia.2014.0009. Epub 2014 May 6. PMID 24801544

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-loop Insulin Delivery: glucose sensor and insulin pump
Period: Overall Study
Arm/Group | Closed-loop Insulin Delivery | Open-loop Insulin Delivery
Started | 8 | 6
Completed | 6 | 6
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-loop Insulin Delivery: standard insulin pump therapy
- Total: Total of all reporting groups
Arm/Group | Closed-loop Insulin Delivery | Open-loop Insulin Delivery | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10) | 45 (10) | 45 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
HbA1c [Mean (Standard Deviation); unit: percentage] | 7.4 (0.7) | 7.4 (0.7) | 7.4 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Time in Euglycaemia
Description: Interstitial blood glucose will be measured every 5 minutes and venous blood glucose every 15 minutes during subject visits 3, 4 and 5 when insulin is being delivered using the closed-loop insulin delivery system. The % time in euglycaemia is to be calculated using these blood glucose values.
Time Frame: 18 months
Measure: Number; unit: percentage of time
Groups:
- Open-loop Insulin Delivery: sensor augmented pump therapy
Arm/Group | Closed-loop Insulin Delivery | Open-loop Insulin Delivery
Number analyzed (Participants) | 8 | 6
percentage of time | 71 | 66.9

2. Secondary Outcome: % Time in Hypoglycaemia
Description: Interstitial blood glucose will be measured every 5 minutes and venous blood glucose every 15 minutes during subject visits 3, 4 and 5 when insulin is being delivered using the closed-loop insulin delivery system. The % time in hypoglycaemia is to be calculated using these blood glucose values.
Time Frame: 18 months
Reporting Status: Not Posted

3. Secondary Outcome: % Time Spent in Hyperglycaemia
Description: Interstitial blood glucose will be measured every 5 minutes and venous blood glucose every 15 minutes during patient visits 3, 4 and 5 when insulin is being delivered using the closed-loop insulin delivery system. The % time in euglycaemia is to be calculated using these blood glucose values.
Time Frame: 18 months
Reporting Status: Not Posted

4. Secondary Outcome: Glycaemic Variability as Measured by MAGE and SD
Description: Glycaemic variability as measured by MAGE and SD Calculation using CGM data
Time Frame: 18 months
Reporting Status: Not Posted

5. Secondary Outcome: Glycaemic Risk as Measured by LBGI and HBG
Description: Glycaemic risk as measured by LBGI and HBG Calculation using CGM data
Time Frame: 18 months
Reporting Status: Not Posted

6. Secondary Outcome: Closed Loop Error Grid Analysis
Description: Closed loop error grid analysis Calculation using CGM data
Time Frame: 18 months
Reporting Status: Not Posted

7. Secondary Outcome: Glucose Area Under the Curve
Description: Glucose area under the curve Calculation using CGM data
Time Frame: 18 months
Reporting Status: Not Posted

8. Secondary Outcome: Insulin Requirement in Units/kg/hr
Description: Calculation using average insulin delivered per hour and bodyweight
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Groups:
- Open-loop: sensor augmented pump
Arm/Group | Closed-loop Insulin Delivery | Open-loop
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes